CLINICAL TRIAL: NCT02587221
Title: A Phase III, Randomized, Observer-Blind, Controlled, Multicenter Clinical Study to Evaluate the Efficacy, Safety and Immunogenicity of an MF59-Adjuvanted Quadrivalent Influenza Vaccine Compared to Non-influenza Vaccine Comparator in Adults ≥ 65 Years of Age
Brief Title: Clinical Study to Evaluate the Efficacy, Safety and Immunogenicity of an MF59-Adjuvanted Quadrivalent Influenza Vaccine Compared to Non-influenza Vaccine Comparator in Adults ≥ 65 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V118_18; 2015-000728-27 (EudraCT Number)
Record Dates: First submitted 2015-10-15; First posted 2015-10-27 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Boostrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aQIV (Experimental): MF59-adjuvanted Quadrivalent Influenza Vaccine (aQIV)
  Interventions: Biological: MF59-adjuvanted Quadrivalent Subunit Inactivated Egg-derived Influenza Vaccine (aQIV)
- Non-influenza Comparator Vaccine (Placebo Comparator): Non-influenza comparator vaccine
  Interventions: Biological: Non-Influenza Comparator (Boostrix)

INTERVENTIONS:
Biological: MF59-adjuvanted Quadrivalent Subunit Inactivated Egg-derived Influenza Vaccine (aQIV) — 1 dose approximately 0.5 mL of aQIV
  Arms: aQIV
Biological: Non-Influenza Comparator (Boostrix) — 1 dose approximately 0.5 mL dose of Non-influenza comparator vaccine (Boostrix)
  Arms: Non-influenza Comparator Vaccine

SUMMARY:
A Phase III, Randomized, Observer-Blind, Controlled, Multicenter Clinical Study to Evaluate the Efficacy, Safety and Immunogenicity of an MF59-Adjuvanted Quadrivalent Influenza Vaccine Compared to Non-influenza Vaccine Comparator in Adults ≥ 65 Years of Age.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 65 years old who are healthy or have co-morbidities
2. Individuals who or whose legal guardian have voluntarily given written consent after the nature of the study has been explained according to local regulatory requirements, prior to study entry.
3. Ability to attend all scheduled visits and to comply with study procedures

Exclusion Criteria:

1. Hypersensitivity, including allergy to any component of vaccines foreseen in this study
2. Abnormal function of the immune system.
3. Receipt of any influenza vaccine within 6 months prior to enrolment in this study or who plan to receive influenza vaccine while participating in the study.
4. Additional eligibility criteria may be discussed by contacting the site

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 6790 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2018-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Program Manager, Study Director — Seqirus
Locations (89):
- Bulgaria (11):
  - MHAT St. Ekaterina, Dimitrovgrad
  - MHAT Sv Nikolay Chudotvoretz Lom, Lom
  - MBAL TRIMONCIUM (Synexus), Plovdiv
  - SHATPPD-Ruse, Rousse
  - Mhat Silistra, Silistra
  - Mc Smolyan, Smolyan
  - Mc Avicena Sofia, Sofia
  - Medical Center Excelsior, Sofia
  - Medical center Synexus Sofia EOOD, Sofia
  - SHATPPD-Sofia, City, Sofia
  - Medical Centre Orpheus OOD (Synexus), Stara Zagora
- Colombia (7):
  - Hospital General de Medellín-Luz Castro de Gutiérrez - E.S.E, Medellín, Antioquia
  - Caja de Compesanción Familiar CAFAM, Bogotá, Cundinamarca
  - Fundacion Cardiomet CEQUIN - Internal Medicine, Armenia
  - Clinica de la Costa, Barranquilla
  - Centro de Atención e Investigación Médica S.A.S. - CAIMED S.A.S., Bogotá
  - Medplus Medicina Prepagada, Bogotá
  - Asociacion IPS Medicos Internistas de Caldas, Manizales
- Czechia (5):
  - CCBR Czech Brno, s.r.o., Brno
  - Centrum ockovani a cestovni mediciny, Hradec Králové
  - FN Hradec Kralove, Hradec Králové
  - CCBR Ostrava, s.r.o., Ostrava
  - CCBR Czech, a.s., Pardubice
- Estonia (6):
  - Center for Clinical and Basic Research, Tallinn, Harju
  - Medicum AS, Tallinn, Harju
  - Merelahe Family Doctors Centre, Tallinn, Harju
  - Vee Family Doctors Centre, Paide, Järvamaa
  - Clinical Research Center, Tartu, Tartu
  - Family Doctors Pullerits & Gavronski, Tartu, Tartu
- Latvia (4):
  - Practice Dr Liga Kozlovska, Balvi
  - Practice Dr Ruta Eglite, Kuldīga
  - Family Doctor Andra Lasmane clinic "ALMA", Riga
  - Practice Dr Inese Petrova, Tukums
- Lithuania (7):
  - JSC Saules seimos medicinos centras, Kaunas
  - Kauno klinikine ligonine, Kaunas
  - Lietuvos Sveikatos Mokslų Universitetas, Kaunas
  - UAB InMedica, Kaunas
  - Klaipeda University Hospital, Klaipėda
  - Republican Siauliai Hospital, Šiauliai
  - CCBR, Vilnius
- Malaysia (8):
  - Hospital Sultanah Bahiyah, Alor Star
  - Hospital Selayang, Batu Caves
  - Klinik Kesihatan Greentown, Ipoh
  - Hospital Raja Perempuan Zainab II, Kota Bharu
  - University Malaya Medical Centre (UMMC), Kuala Lumpur
  - Klinik Kesihatan Seremban 2, Seremban
  - Hospital Seri Manjung, Seri Manjung
  - Hospital Sibu, Sibu
- Philippines (6):
  - De La Salle Health Sciences Institute, Dasmariñas, Cavite
  - West Visayas State University - Medical Center, Jaro, Iloilo
  - Quirino Memorial Medical Center, Quezon City, National Capital Region
  - Marilao St. Michael Family Hospital, Bulacan
  - Philippine General Hospital, Manila
  - San Juan De Dios Hospital, Pasay
- Poland (15):
  - Synexus Polska Sp. z o.o, Poznan, Greater Poland Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej VITAMED, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Synexus Polska Sp. z o.o., Wroclaw, Lower Silesian Voivodeship
  - NZOZ Centrum Medyczne "OMEGA" sp. z o.o., Płock, Masovian Voivodeship
  - Centrum Medyczne Pratia Warszawa, Warsaw, Masovian Voivodeship
  - Specjalistyczny Osrodek Medycyny Wieku Dojrzalego, Warsaw, Masovian Voivodeship
  - Synexus Polska Sp. z o.o., Gdansk, Pomeranian Voivodeship
  - Centrum Medyczne Pratia Gdynia, Gdynia, Pomeranian Voivodeship
  - Centrum Medyczne Pratia Katowice, Katowice, Silesian Voivodeship
  - Praktyka Lekarzy Rodzinnych SALUS, Katowice, Silesian Voivodeship
  - Centrum Medyczne PRATIA Bydgoszcz, Bydgoszcz
  - Specjalistyczny Osrodek Medycyny Wieku Dojrzalego sp. z o.o., Lodz
  - RCMed Oddział Nowy Duninow, Nowy Duninów
  - RCMed Oddzial Sochaczew, Sochaczew
  - Medical Trials Institute, Torun
- Romania (8):
  - Cabinet dr. Dana OLAR, Arad
  - Centrul Medical de Diagnostic si Tratament Ambulator NEOMED, Brasov
  - Cabinet Medical Individual Craciun-Nicodin Maria Marcela, Bucharest
  - Centrul Medical Sana, Bucharest
  - Clinica Medicala Synexus, Bucharest
  - Spitalul Clinic C.F. Cluj-Napoca, Cluj-Napoca
  - Clintrial Medical Center, Reșca
  - Fundatia Cardioprevent, Timișoara
- Thailand (4):
  - Ramathibodi Hospital, Bangkok
  - Mahidol University (MU) - Faculty of Tropical Medicine, Bangkok
  - Khon Kaen University - Srinagarind Hospital - Medicine, Khon Kaen
  - Bamrasnaradura Infectious Diseases Institute (BIDI), Nonthaburi
- Turkey (Türkiye) (8):
  - Ankara Training and Research Hospital, Ankara
  - Hacettepe University Medical Faculty, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Istanbul University Cerrahpasa Medical Faculty, Cerrahpaşa
  - Ataturk University Medical Faculty, Erzurum
  - Ege University Medical Faculty, Izmir
  - Kocaeli University Research and Application Hospital, Kocaeli
  - Sakarya Training and Research Hospital, Sakarya

REFERENCES:
- [Derived] Beran J, Reynales H, Poder A, Yu CY, Pitisuttithum P, Yuan LL, Vermeulen W, Verhoeven C, Leav B, Zhang B, Sawlwin D, Hamers-Heijnen E, Edelman J, Smolenov I. Prevention of influenza during mismatched seasons in older adults with an MF59-adjuvanted quadrivalent influenza vaccine: a randomised, controlled, multicentre, phase 3 efficacy study. Lancet Infect Dis. 2021 Jul;21(7):1027-1037. doi: 10.1016/S1473-3099(20)30694-0. Epub 2021 Feb 9. PMID 33577767

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled male and female adults ≥ 65 years old who were healthy or had co-morbidities.
Pre-assignment Details: Screening criteria applied.
Groups:
- aQIV: A single dose of approximately 0.5 mL of aQIV was administered on Day 1.
- Non-influenza Comparator Vaccine: A single dose of approximately 0.5 mL dose of Boostrix was administered on Day 1. (Boostrix = Non-influenza comparator vaccine)
Period: Overall Study
Arm/Group | aQIV | Non-influenza Comparator Vaccine
Started | 3394 | 3396
Treated | 3379 | 3382
Completed | 3263 | 3273
Not Completed | 131 | 123
Not completed — Adverse Event | 3 | 3
Not completed — Death | 33 | 34
Not completed — Withdrawal by Subject | 66 | 61
Not completed — Lost to Follow-up | 21 | 19
Not completed — Protocol Violation | 6 | 5
Not completed — Other Reason or Unspecified | 2 | 1

BASELINE CHARACTERISTICS:
Population: Total Number of Subjects Enrolled
Groups:
- aQIV: Subjects received one dose of aQIV vaccine
- Non-influenza Comparator Vaccine: Subjects received one dose of non-influenza comparator vaccine (Boostrix)
- Total: Total of all reporting groups
Arm/Group | aQIV | Non-influenza Comparator Vaccine | Total
Number analyzed (Participants) | 3394 | 3396 | 6790
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (5.53) | 71.8 (5.36) | 71.9 (5.44)
Age, Customized [Count of Participants; unit: Participants]
  65 to 74 years | 2416 | 2406 | 4822
  75 to 84 years | 893 | 928 | 1821
  . 85 years | 85 | 62 | 147
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2105 | 2089 | 4194
  Male | 1289 | 1307 | 2596
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 615 | 607 | 1222
  Not Hispanic or Latino | 2773 | 2779 | 5552
  Unknown or Not Reported | 6 | 10 | 16
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 62 | 59 | 121
  Asian | 1139 | 1159 | 2298
  Black or African American | 1 | 0 | 1
  White | 1642 | 1629 | 3271
  Other | 550 | 549 | 1099
Region of Enrollment [Number; unit: participants]
  Bulgaria | 183 | 183 | 366
  Colombia | 613 | 611 | 1224
  Czechia | 182 | 184 | 366
  Estonia | 324 | 317 | 641
  Latvia | 142 | 140 | 282
  Lithuania | 223 | 224 | 447
  Malaysia | 446 | 453 | 899
  Philippines | 453 | 457 | 910
  Poland | 361 | 358 | 719
  Romania | 180 | 176 | 356
  Thailand | 242 | 248 | 490
  Turkey | 45 | 45 | 90
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: According to data availability.
  kg/m^2
    number analyzed (Participants) | 3391 | 3393 | 6784
    (all) | 27.05 (4.989) | 26.96 (4.995) | 27.00 (4.992)
Previous Seasonal Influenza Vaccine in the Past 5 Years [Count of Participants; unit: Participants]
  Yes | 991 | 1021 | 2012
  No | 2403 | 2375 | 4778
Comorbidity Score [Count of Participants; unit: Participants] — Comorbidity risk scores were assessed among other baseline characteristics as a validated predictor of risk of influenza complications in subjects ≥65 years of age using a model-based approach assessing 5 disease classifications (pulmonary disease, heart disease, renal disease, dementia or stroke, and non-hematological and hematological cancer [excluding cancer of the skin other than melanoma]). Using this model, a score of <50 was considered low risk and a score of ≥50 was considered high risk for hospitalization due to pneumonia or influenza and death from any cause.
  Participants
    < 50 | 2472 | 2474 | 4946
    ≥ 50 | 922 | 922 | 1844
Smoking Status [Count of Participants; unit: Participants]
  Smoking | 325 | 335 | 660
  Not smoking | 3069 | 3061 | 6130

OUTCOME MEASURES:

1. Primary Outcome: Absolute Vaccine Efficacy (VE) of aQIV Versus Non-influenza Comparator Based on RT-PCR-confirmed Influenza Due to Any Strain Using Protocol Defined ILI Definition.
Description: The primary efficacy endpoint was the time of first-occurrence of RT-PCR-confirmed influenza due to any strain of influenza regardless of antigenic match to the strains selected for the seasonal vaccine from Day 21 through 180 days after vaccination or end of the influenza season, whichever is longer, using protocol defined ILI definition. Absolute vaccine efficacy is VE=1-HR, where HR is the hazard ratio of aQIV vs non-influenza comparator estimated by the Cox proportional hazards model for the primary endpoint.
Time Frame: Day 21 to Day 180 after vaccination or end of influenza season, whichever is longer
Population: The Full Analysis Set (FAS) Efficacy, consisting of all randomized subjects who received a study treatment, were under observation for at least 21 days post-vaccination and provided efficacy data, was used for analysis
Measure: Number; unit: Number of cases
Arm/Group | aQIV | Non-influenza Comparator Vaccine
Number analyzed (Participants) | 3368 | 3372
Number of cases | 122 | 151
Statistical Analysis 1: Comparison: aQIV vs Non-influenza Comparator Vaccine; The efficacy of aQIV would be demonstrated if the LL of the two-sided multiplicity adjusted 95%CI for the vaccine efficacy is >40%; Test type: Other — VE=1-HR, where HR is the hazard ratio estimated by the Cox proportional hazards model for time to first occurrence of RT-PCR confirmed due to any strain. An ILI was defined as presence of ≥1 respiratory symptom (e.g. sore throat, cough, sputum production, wheezing, or difficulty breathing) concurrently with ≥1 systemic symptom (temp >37.2°C/99°F, chills, tiredness, headache, or myalgia) (protocol defined ILI definition); Regression, Cox; Adjusted for covariates; Vaccine efficacy (VE) = 19.80, 97.45% CI 2-sided [-5.27 to 38.91]

2. Primary Outcome: Safety Endpoint: The Percentage of Subjects in the Solicited Safety Subset With Solicited Local and Systemic Adverse Events (AE)
Description: Safety of vaccination was assessed in terms of percentage of subjects reporting solicited local and systemic AEs up to 7 days after vaccination.
Time Frame: Day 1 through Day 7
Population: SOLICITED SAFETY SET = randomly selected subset of all treated subjects, with solicited safety assessments beyond 30 minutes
Measure: Number; unit: Percentage of subjects
Arm/Group | aQIV | Non-influenza Comparator Vaccine
Number analyzed (Participants) | 665 | 667
Percentage of subjects
  Any solicited AE | 34.3 | 32.2
  Any local solicited AE | 24.4 | 19.6
  Any systemic solicited AE | 19.2 | 16.3
  Other | 6.2 | 3.9

3. Primary Outcome: Safety Endpoint: Percentage of Subjects With Medically-attended Adverse Events (MAAEs)
Description: Safety of vaccination was assessed in terms of percentage of subjects reporting medically attended AEs within 30 days after of first occurrence RT-PCR confirmed influenza.
Time Frame: Within 30 days after of first occurrence RT-PCR confirmed Influenza
Population: UNSOLICITED SAFETY SET - consisting of treated subjects with unsolicited AE data was used for analysis.
Measure: Number; unit: Percentage of subjects
Arm/Group | aQIV | Non-influenza Comparator Vaccine
Number analyzed (Participants) | 3368 | 3372
Percentage of subjects | 0.7 | 0.4

4. Primary Outcome: Safety Endpoint: Percentages of Subjects With Any Unsolicited AE
Description: Safety of vaccination was assessed in terms of percentage of subjects reporting unsolicited AEs up to 21 days after vaccination.
Time Frame: Day 1 through Day 366
Population: UNSOLICITED SAFETY SET - treated subjects with unsolicited AE data was used for analysis.
Measure: Number; unit: Percentage of subjects
Arm/Group | aQIV | Non-influenza Comparator Vaccine
Number analyzed (Participants) | 3380 | 3377
Percentage of subjects | 21.5 | 21.2

5. Primary Outcome: Safety Endpoint: Percentages of Subjects With Serious Adverse Events (SAE), AEs Leading to Withdrawal, New Onset of Chronic Disease (NOCD), and Adverse Events of Special Interest (AESI)
Description: Safety of vaccination was assessed in terms of percentage of subjects reporting SAEs, AEs leading to withdrawal, NOCDs, and AESIs up to 366 days after vaccination.
Time Frame: Day 1 to Day 366
Population: UNSOLICITED SAFETY SET - treated subjects with unsolicited AE data was used for analysis.
Measure: Number; unit: Percentage of subjects
Arm/Group | aQIV | Non-influenza Comparator Vaccine
Number analyzed (Participants) | 3380 | 3377
Percentage of subjects
  Any unsolicited SAE | 7.0 | 6.9
  Any related SAE | 0.0 | 0.0
  Any unsolicited AEs leading to withdrawal | 1.1 | 1.1
  Any NOCD | 9.5 | 9.0
  Any AESI | 0.1 | 0.2

6. Secondary Outcome: Absolute Vaccine Efficacy (VE) of aQIV Versus Non-influenza Comparator Based on RT-PCR-confirmed Influenza Due to Any Strain Using Modified CDC ILI Definition.
Description: The secondary efficacy endpoint was the time of first-occurrence of RT-PCR-confirmed influenza due to any strain of influenza regardless of antigenic match to the strains selected for the seasonal vaccine from Day 21 through 180 days after vaccination or end of the influenza season, whichever is longer, using modified CDC ILI definition. Absolute vaccine efficacy is VE=1-HR, where HR is the hazard ratio of aQIV vs non-influenza comparator estimated by the Cox proportional hazards model for the secondary efficacy endpoint.
Time Frame: Day 21 to Day 180 after vaccination or end of influenza season, whichever is longer
Population: as for outcome 1
Measure: Number; unit: Number of cases
Arm/Group | aQIV | Non-influenza Comparator Vaccine
Number analyzed (Participants) | 3368 | 3372
Number of cases | 83 | 121
Statistical Analysis 1: Comparison: aQIV vs Non-influenza Comparator Vaccine; Test type: Other — VE=1-HR, where HR is the hazard ratio estimated by the Cox proportional hazards model for time to first occurrence of RT-PCR confirmed due to any strain. An ILI was defined as the presence of fever (temperature >37.2°C) with cough or sore throat (modified CDC ILI definition); Regression, Cox; Adjusted for covariates; Vaccine efficacy (VE) = 32.12, 95% CI 2-sided [10.23 to 48.67]

7. Secondary Outcome: Absolute Vaccine Efficacy (VE) of aQIV Versus Non-influenza Comparator Based on Culture Confirmed Influenza Due to Any Strain of Influenza Antigenically Matched to the Strains Selected for the Seasonal Vaccine Using Protocol Defined ILI Definition.
Description: The secondary efficacy endpoint was the time of first-occurrence of culture confirmed influenza due to any strain of influenza antigenically matched to the strains selected for the seasonal vaccine from Day 21 through 180 days after vaccination or end of the influenza season, whichever is longer, using protocol defined ILI definition. Absolute vaccine efficacy is VE=1-HR, where HR is the hazard ratio of aQIV vs non-influenza comparator estimated by the Cox proportional hazards model for the secondary endpoint.
Time Frame: Day 21 to Day 180 after vaccination or end of influenza season, whichever is longer
Population: as for outcome 1
Measure: Number; unit: Number of cases
Arm/Group | aQIV | Non-influenza Comparator Vaccine
Number analyzed (Participants) | 3368 | 3372
Number of cases | 7 | 14
Statistical Analysis 1: Comparison: aQIV vs Non-influenza Comparator Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Other — VE=1-HR, where HR is the hazard ratio estimated by the Cox proportional hazards model for time to first occurrence of culture confirmed influenza due to any strain of influenza antigenically matched to the vaccine strains. An ILI was defined as the presence of ≥1 respiratory symptom (eg. sore throat, cough, sputum production, wheezing, or difficulty breathing) concurrently with ≥1 systemic symptom (temp >37.2°C/99°F, chills, tiredness, headache, or myalgia) (protocol defined ILI definition); Regression, Cox; Adjusted for covariates; Vaccine efficacy (VE) = 49.94, 95% CI 2-sided [-24.03 to 79.79]

8. Secondary Outcome: Absolute Vaccine Efficacy (VE) of aQIV Versus Non-influenza Comparator Based on Culture Confirmed Influenza Due to Any Strain of Influenza Antigenically Matched to the Strains Selected for the Seasonal Vaccine Using Modified CDC ILI Definition.
Description: The secondary efficacy endpoint was the time of first-occurrence of culture confirmed influenza due to any strain of influenza antigenically matched to the strains selected for the seasonal vaccine from Day 21 through 180 days after vaccination or end of the influenza season, whichever is longer, using modified CDC ILI definition. Absolute vaccine efficacy is VE=1-HR, where HR is the hazard ratio of aQIV vs non-influenza comparator estimated by the Cox proportional hazards model for the secondary endpoint.
Time Frame: Day 21 to Day 180 after vaccination or end of influenza season, whichever is longer
Population: as for outcome 1
Measure: Number; unit: Number of cases
Arm/Group | aQIV | Non-influenza Comparator Vaccine
Number analyzed (Participants) | 3368 | 3372
Number of cases | 5 | 13
Statistical Analysis 1: Comparison: aQIV vs Non-influenza Comparator Vaccine; Test type: Other — VE=1-HR, where HR is the hazard ratio estimated by the Cox proportional hazards model for time to first occurrence of culture confirmed influenza due to any strain of influenza antigenically matched to the strains selected for the seasonal vaccine. An ILI was defined as presence of fever (temperature >37.2°C) with cough or sore throat (modified CDC ILI definition); Regression, Cox; Adjusted for covariates; Vaccine efficacy (VE) = 61.50, 95% CI 2-sided [-7.98 to 86.28]

9. Secondary Outcome: Absolute Vaccine Efficacy (VE) of aQIV Versus Non-influenza Comparator Based on Culture Confirmed Influenza Due to Any Strain of Influenza Regardless of Antigenic Match Using Protocol Defined ILI Definition.
Description: The secondary efficacy endpoint was the time of first-occurrence of culture confirmed influenza due to any strain of influenza regardless of antigenic match from Day 21 through 180 days after vaccination or end of the influenza season, whichever is longer, using protocol defined ILI definition. Absolute vaccine efficacy is VE=1-HR, where HR is the hazard ratio of aQIV vs non-influenza comparator estimated by the Cox proportional hazards model for the secondary endpoint.
Time Frame: Day 21 to Day 180 after vaccination or end of influenza season, whichever is longer
Population: as for outcome 1
Measure: Number; unit: Number of cases
Arm/Group | aQIV | Non-influenza Comparator Vaccine
Number analyzed (Participants) | 3368 | 3372
Number of cases | 58 | 81
Statistical Analysis 1: Comparison: aQIV vs Non-influenza Comparator Vaccine; Test type: Other — VE=1-HR, where HR is the hazard ratio estimated by the Cox proportional hazards model for time to first occurrence of culture confirmed influenza due to any vaccine strain regardless of antigenic match. An ILI was defined as the presence of ≥1 respiratory symptom (e.g. sore throat, cough, sputum production, wheezing, or difficulty breathing) concurrently with ≥1 systemic symptom (temp >37.2°C/99°F, chills, tiredness, headache, or myalgia) (protocol defined ILI definition); Regression, Cox; Adjusted for covariates; Vaccine efficacy (VE) = 28.66, 95% CI 2-sided [0.05 to 49.08]

10. Secondary Outcome: Absolute Vaccine Efficacy (VE) of aQIV Versus Non-influenza Comparator Based on Culture Confirmed Influenza Due to Any Strain of Influenza Regardless of Antigenic Match Using Modified CDC ILI Definition.
Description: The secondary efficacy endpoint was the time of first-occurrence of culture confirmed influenza due to any strain of influenza regardless of antigenic match from Day 21 through 180 days after vaccination or end of the influenza season, whichever is longer, using modified CDC ILI definition. Absolute vaccine efficacy is VE=1-HR, where HR is the hazard ratio of aQIV vs non-influenza comparator estimated by the Cox proportional hazards model for the secondary endpoint.
Time Frame: Day 7 to Day 180 after vaccination or end of influenza season, whichever is longer
Population: as for outcome 1
Measure: Number; unit: Number of cases
Arm/Group | aQIV | Non-influenza Comparator Vaccine
Number analyzed (Participants) | 3368 | 3372
Number of cases | 44 | 66
Statistical Analysis 1: Comparison: aQIV vs Non-influenza Comparator Vaccine; Test type: Other — VE=1-HR, where HR is the hazard ratio estimated by the Cox proportional hazards model for time to first occurrence of culture confirmed influenza due to any strain of influenza regardless of antigenic match An ILI was defined as presence of fever (temperature >37.2°C) with cough or sore throat (modified CDC ILI definition); Regression, Cox; Adjusted for covariates; Vaccine efficacy (VE) = 33.47, 95% CI 2-sided [2.56 to 54.57]

11. Secondary Outcome: Absolute Vaccine Efficacy (VE) of aQIV Versus Non-influenza Comparator Based on Culture Confirmed Influenza Due to Any Strain of Influenza Antigenically Unmatched to the Strains Selected for the Seasonal Vaccine Using Protocol Defined ILI Definition.
Description: The secondary efficacy endpoint was the time of first-occurrence of culture confirmed influenza due to any strain of influenza antigenically unmatched to the strains selected for the seasonal vaccine from Day 21 through 180 days after vaccination or end of the influenza season, whichever is longer, using protocol defined ILI definition. Absolute vaccine efficacy is VE=1-HR, where HR is the hazard ratio of aQIV vs non-influenza comparator estimated by the Cox proportional hazards model for the secondary endpoint.
Time Frame: Day 21 to Day 180 after vaccination or end of influenza season, whichever is longer
Population: as for outcome 1
Measure: Number; unit: Number of cases
Arm/Group | aQIV | Non-influenza Comparator Vaccine
Number analyzed (Participants) | 3368 | 3372
Number of cases | 51 | 67
Statistical Analysis 1: Comparison: aQIV vs Non-influenza Comparator Vaccine; Test type: Other — VE=1-HR, where HR is the hazard ratio estimated by the Cox proportional hazards model for time to first occurrence of culture confirmed influenza due to any strain of influenza antigenically unmatched to the vaccine strains. An ILI is the presence of ≥1 respiratory symptom (e.g. sore throat, cough, sputum production, wheezing, or difficulty breathing) concurrently with ≥1 systemic symptom (temp >37.2°C/99°F, chills, tiredness, headache, or myalgia) (protocol defined ILI definition); Regression, Cox; Adjusted for covariates; Vaccine efficacy (VE) = 23.79, 95% CI 2-sided [-9.69 to 47.05]

12. Secondary Outcome: Absolute Vaccine Efficacy (VE) of aQIV Versus Non-influenza Comparator Based on Culture Confirmed Influenza Due to Any Strain of Influenza Antigenically Unmatched to the Strains Selected for the Seasonal Vaccine Using Modified CDC ILI Definition.
Description: The secondary efficacy endpoint was the time of first-occurrence of culture confirmed influenza due to any strain of influenza antigenically unmatched to the strains selected for the seasonal vaccine from Day 21 through 180 days after vaccination or end of the influenza season, whichever is longer, using modified CDC ILI definition. Absolute vaccine efficacy is VE=1-HR, where HR is the hazard ratio of aQIV vs non-influenza comparator estimated by the Cox proportional hazards model for the secondary endpoint.
Time Frame: Day 21 to Day 180 after vaccination or end of influenza season, whichever is longer
Population: as for outcome 1
Measure: Number; unit: Number of cases
Arm/Group | aQIV | Non-influenza Comparator Vaccine
Number analyzed (Participants) | 3368 | 3372
Number of cases | 39 | 53
Statistical Analysis 1: Comparison: aQIV vs Non-influenza Comparator Vaccine; Test type: Other — VE=1-HR, where HR is the hazard ratio estimated by the Cox proportional hazards model for time to first occurrence of culture confirmed influenza due to any strain of influenza antigenically unmatched to the strains selected for the seasonal vaccine. An ILI was defined as presence of fever (temperature >37.2°C) with cough or sore throat (modified CDC ILI definition); Regression, Cox; Adjusted for covariates; Vaccine efficacy (VE) = 26.11, 95% CI 2-sided [-11.71 to 51.13]

13. Secondary Outcome: Immunogenicity Endpoint: Geometric Mean Hemagglutination Inhibition (HI) Titers (GMT)
Description: The log-transformed antibody titers (GMT) at Day 1 and Day 22 were evaluated using an analysis of covariance (ANCOVA) model including factors for site/country, pre-vaccination titer, age, and comorbidity.
Time Frame: Days 1 and 22
Population: The FAS Immunogenicity, consisting of all randomized subjects who received a study treatment, and provided immunogenicity data at Days 1 and 22, was used for analysis
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | aQIV | Non-influenza Comparator Vaccine
Number analyzed (Participants) | 1324 | 332
titer
  A/H1N1 Day 1 | 31.86 [28.49 to 35.63] | 36.19 [30.05 to 43.57]
  A/H1N1 Day 22 | 438.79 [403.82 to 476.79] | 29.43 [25.63 to 33.79]
  A/H3N2 Day 1 | 28.31 [25.43 to 31.52] | 27.56 [23.05 to 32.95]
  A/H3N2 Day 22 | 572.80 [525.08 to 624.86] | 27.06 [23.42 to 31.25]
  B/Yamagata Day 1 | 13.83 [12.81 to 14.92] | 13.13 [11.57 to 14.91]
  B/Yamagata Day 22 | 86.77 [79.94 to 94.19] | 12.49 [10.90 to 14.30]
  B/Victoria Day 1 | 12.77 [11.81 to 13.81] | 12.26 [10.77 to 13.96]
  B/Victoria Day 22 | 104.26 [95.77 to 113.50] | 11.25 [9.77 to 12.94]

14. Secondary Outcome: Immunogenicity Endpoint: Geometric Mean Ratio (GMR) of Post-vaccination HI Titer Over the Pre-vaccination HI Titer
Description: The GMR was assessed as the postvaccination HI titer divided by the prevaccination HI titer (Day 22/Day 1).
Time Frame: Day 22/Day 1
Population: The FAS Immunogenicity, consisting of all randomized subjects who received a study treatment, and provided immunogenicity data at Days 1 and 22, was used for analysis GMR B/Vic: 0.94 to )
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | aQIV | Non-influenza Comparator Vaccine
Number analyzed (Participants) | 1324 | 332
ratio
  A/H1N1 | 14.17 [12.84 to 15.64] | 0.89 [0.76 to 1.05]
  A/H3N2 | 22.65 [20.48 to 25.06] | 1.08 [0.92 to 1.28]
  B/Yamagata | 6.58 [6.02 to 7.20] | 0.97 [0.84 to 1.13]
  B/Victoria | 8.59 [7.83 to 9.42] | 0.94 [0.81 to 1.10]

15. Secondary Outcome: Immunogenicity Endpoint: Percentages of Subjects With an HI Titer ≥1:40
Description: The percentage of subjects vaccinated with aQIV with a HI antibody titers ≥1:40 was assessed for each of the 4 strains Assessment criteria was considered fulfilled if the lower bound of the two-sided 95% CI for percent of subjects with HI antibody titer ≥1:40 met or exceeded 60% at Day 22.
Time Frame: Day 22
Population: as for outcome 13
Measure: Mean (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aQIV | Non-influenza Comparator Vaccine
Number analyzed (Participants) | 1324 | 332
Percentage of subjects
  A/H1N1 | 96.2 [95.05 to 97.18] | 46.7 [41.18 to 52.21]
  A/H3N2 | 95.6 [94.37 to 96.66] | 41.7 [36.32 to 47.21]
  B/Yamagata | 79.2 [76.95 to 81.40] | 21.5 [17.20 to 26.35]
  B/Victoria | 81.6 [79.39 to 83.65] | 18.4 [14.40 to 23.03]

16. Secondary Outcome: Immunogenicity Endpoint: Percentages of Subjects Who Achieved Seroconversion (SCR)
Description: The percentage of subjects achieving SCR at Day 22 was assessed for each of the 4 strains. SCR is defined as HI titer ≥1:40 for subjects seronegative at baseline (HI titer <1:10) or a minimum 4-fold increase in HI titer for subjects seropositive at baseline (HI titer ≥1:10) on Day 22. Assessment criteria was considered fulfilled if the lower bound of the two-sided 95% CI for the percentage of subjects achieving an HI antibody SCR met or exceeded 30% at Day 22.
Time Frame: Day 22
Population: analysis.
Measure: Mean (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aQIV | Non-influenza Comparator Vaccine
Number analyzed (Participants) | 1324 | 332
Percentage of subjects
  A/H1N1 | 78.0 [75.66 to 80.21] | 2.1 [0.85 to 4.31]
  A/H3N2 | 84.6 [82.52 to 86.49] | 3.9 [2.11 to 6.62]
  B/Yamagata | 60.8 [58.06 to 63.41] | 3.6 [1.89 to 6.27]
  B/Victoria | 65.5 [62.88 to 68.10] | 2.1 [0.85 to 4.31]

17. Post Hoc Outcome: Absolute Vaccine Efficacy (VE) of aQIV Versus Non-influenza Comparator Based on RT-PCR-confirmed Influenza Due to Any Strain Using WHO ILI Definition.
Description: The post-hoc efficacy endpoint was the time of first-occurrence of RT-PCR-confirmed influenza due to any strain of influenza regardless of antigenic match to the strains selected for the seasonal vaccine from Day 21 through 180 days after vaccination or end of the influenza season, whichever is longer, using WHO ILI definition. Absolute vaccine efficacy is VE=1-HR, where HR is the hazard ratio of aQIV vs non-influenza comparator estimated by the Cox proportional hazards model for the post-hoc efficacy endpoint
Time Frame: Day 21 to Day 180 after vaccination or end of influenza season, whichever is longer
Population: as for outcome 1
Measure: Number; unit: Number of cases
Arm/Group | aQIV | Non-influenza Comparator Vaccine
Number analyzed (Participants) | 3368 | 3372
Number of cases | 39 | 79
Statistical Analysis 1: Comparison: aQIV vs Non-influenza Comparator Vaccine; Test type: Other — VE=1-HR, where HR is the hazard ratio estimated by the Cox proportional hazards model for time to first occurrence of RT-PCR confirmed due to any strain. An ILI was defined as presence of fever (temperature ≥38°C) with cough (WHO ILI definition); Regression, Cox; Adjusted for covariates; Vaccine efficacy (VE) = 51.08, 95% CI 2-sided [28.21 to 66.67]

18. Post Hoc Outcome: Absolute Vaccine Efficacy (VE) of aQIV Versus Non-influenza Comparator Based on Culture Confirmed Influenza Due to Any Strain of Influenza Antigenically Matched to the Strains Selected for the Seasonal Vaccine Using WHO ILI Definition.
Description: The post-hoc efficacy endpoint was the time of first-occurrence of culture confirmed influenza due to any strain of influenza antigenically matched to the strains selected for the seasonal vaccine from Day 21 through 180 days after vaccination or end of the influenza season, whichever is longer, using WHO ILI definition. Absolute vaccine efficacy is VE=1-HR, where HR is the hazard ratio of aQIV vs non-influenza comparator estimated by the Cox proportional hazards model for the post-hoc endpoint.
Time Frame: Day 21 to Day 180 after vaccination or end of influenza season, whichever is longer
Population: as for outcome 1
Measure: Number; unit: Number of cases
Arm/Group | aQIV | Non-influenza Comparator Vaccine
Number analyzed (Participants) | 3368 | 3372
Number of cases | 2 | 8
Statistical Analysis 1: Comparison: aQIV vs Non-influenza Comparator Vaccine; Test type: Other — VE=1-HR, where HR is the hazard ratio estimated by the Cox proportional hazards model for time to first occurrence of culture confirmed influenza due to any strain of influenza antigenically matched to the strains selected for the seasonal vaccine. An ILI was defined as presence of fever (temperature ≥38°C) with cough (WHO ILI definition); Regression, Cox; Adjusted for covariates; Vaccine efficacy (VE) = 74.96, 95% CI 2-sided [-17.93 to 94.68]

19. Post Hoc Outcome: Absolute Vaccine Efficacy (VE) of aQIV Versus Non-influenza Comparator Based on Culture Confirmed Influenza Due to Any Strain of Influenza Regardless of Antigenic Match Using WHO ILI Definition
Description: The post-hoc efficacy endpoint was the time of first-occurrence of culture confirmed influenza due to any strain of influenza regardless of antigenic match from Day 21 through 180 days after vaccination or end of the influenza season, whichever is longer, using WHO ILI definition. Absolute vaccine efficacy is VE=1-HR, where HR is the hazard ratio of aQIV vs non-influenza comparator estimated by the Cox proportional hazards model for the post-hoc endpoint.
Time Frame: Day 21 to Day 180 after vaccination or end of influenza season, whichever is longer
Population: as for outcome 1
Measure: Number; unit: Number of cases
Arm/Group | aQIV | Non-influenza Comparator Vaccine
Number analyzed (Participants) | 3368 | 3372
Number of cases | 18 | 45
Statistical Analysis 1: Comparison: aQIV vs Non-influenza Comparator Vaccine; Test type: Other — VE=1-HR, where HR is the hazard ratio estimated by the Cox proportional hazards model for time to first occurrence of culture confirmed influenza due to any strain of influenza regardless of antigenic match. An ILI was defined as presence of fever (temperature ≥38°C) with cough (WHO ILI definition); Regression, Cox; Adjusted for covariates; Vaccine efficacy (VE) = 60.17, 95% CI 2-sided [31.19 to 76.94]

20. Post Hoc Outcome: Absolute Vaccine Efficacy (VE) of aQIV Versus Non-influenza Comparator Based on Culture Confirmed Influenza Due to Any Strain of Influenza Antigenically Unmatched to the Strains Selected for the Seasonal Vaccine Using WHO ILI Definition.
Description: The post-hoc efficacy endpoint was the time of first-occurrence of culture confirmed influenza due to any strain of influenza antigenically unmatched to the strains selected for the seasonal vaccine from Day 21 through 180 days after vaccination or end of the influenza season, whichever is longer, using WHO ILI definition. Absolute vaccine efficacy is VE=1-HR, where HR is the hazard ratio of aQIV vs non-influenza comparator estimated by the Cox proportional hazards model for the post-hoc endpoint.
Time Frame: Day 21 to Day 180 after vaccination or end of influenza season, whichever is longer
Population: as for outcome 1
Measure: Number; unit: Number of cases
Arm/Group | aQIV | Non-influenza Comparator Vaccine
Number analyzed (Participants) | 3368 | 3372
Number of cases | 16 | 37
Statistical Analysis 1: Comparison: Non-influenza Comparator Vaccine; Test type: Other — VE=1-HR, where HR is the hazard ratio estimated by the Cox proportional hazards model for time to first occurrence of culture confirmed influenza due to any strain of influenza antigenically unmatched to the strains selected for the seasonal vaccine. An ILI was defined as presence of fever (temperature ≥38°C) with cough (WHO ILI definition); Regression, Cox; Adjusted for covariates; Vaccine efficacy (VE) = 57.02, 95% CI 2-sided [22.73 to 76.09]

ADVERSE EVENTS:
Time Frame: Solicited AEs: Day 1 to Day 7; SAEs: Day 1 to Day 366; and Unsolicited AEs: Day 1 to Day 22.
Groups:
- aQIV: A single dose of approximately 0.5 mL of aQIV was administered on Day 1 (NH 2016/17, SH 2017).
- Non-influenza Comparator Vaccine: Non-influenza Comparator Vaccine / A single dose of approximately 0.5 mL dose of Boostrix was administered on Day 1 (NH 2016/17, SH 2017). (Boostrix = Non-influenza comparator vaccine)
Arm/Group | aQIV | Non-influenza Comparator Vaccine
All-Cause Mortality (participants affected / at risk) | 33/3380 | 34/3377
Serious Adverse Events (participants affected / at risk) | 238/3380 | 234/3377
Other Adverse Events (participants affected / at risk) | 227/665 | 218/667
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | aQIV (N=3380) | Non-influenza Comparator Vaccine (N=3377)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 2
Polycythaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 12 | 19
Atrial fibrillation (Cardiac disorders) | 11 | 10
Angina unstable (Cardiac disorders) | 4 | 7
Cardiac failure (Cardiac disorders) | 6 | 5
Angina pectoris (Cardiac disorders) | 4 | 6
Myocardial infarction (Cardiac disorders) | 4 | 5
Cardiac failure acute (Cardiac disorders) | 3 | 3
Cardiac failure congestive (Cardiac disorders) | 2 | 4
Acute coronary syndrome (Cardiac disorders) | 2 | 3
Cardiac failure chronic (Cardiac disorders) | 1 | 3
Coronary artery disease (Cardiac disorders) | 3 | 1
Cardiac arrest (Cardiac disorders) | 2 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 2
Arrhythmia (Cardiac disorders) | 1 | 1
Atrial flutter (Cardiac disorders) | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Cor pulmonale (Cardiac disorders) | 2 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 2
Mitral valve incompetence (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 2 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Cardiac asthma (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1
Cor pulmonale acute (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 3 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1
Autoimmune thyroiditis (Endocrine disorders) | 1 | 2
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Toxic nodular goitre (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 4 | 4
Angle closure glaucoma (Eye disorders) | 1 | 0
Dacryostenosis acquired (Eye disorders) | 0 | 1
Macular fibrosis (Eye disorders) | 1 | 0
Polypoidal choroidal vasculopathy (Eye disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2
Pancreatitis (Gastrointestinal disorders) | 1 | 2
Pancreatitis acute (Gastrointestinal disorders) | 1 | 2
Chronic gastritis (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Change of bowel habit (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatic cyst (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 7 | 3
Influenza like illness (General disorders) | 0 | 2
Sudden cardiac death (General disorders) | 0 | 2
Medical device pain (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 4
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 2
Cholelithiasis (Hepatobiliary disorders) | 3 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Hepatitis chronic persistent (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Pneumonia (Infections and infestations) | 19 | 18
Urinary tract infection (Infections and infestations) | 6 | 2
Cellulitis (Infections and infestations) | 2 | 5
Gastroenteritis (Infections and infestations) | 4 | 2
Sepsis (Infections and infestations) | 1 | 3
Diabetic foot infection (Infections and infestations) | 3 | 0
Pneumonia bacterial (Infections and infestations) | 2 | 1
Pneumonia klebsiella (Infections and infestations) | 2 | 1
Appendicitis (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 1
Cholecystitis infective (Infections and infestations) | 0 | 2
Dengue fever (Infections and infestations) | 0 | 2
Diverticulitis (Infections and infestations) | 0 | 2
Erysipelas (Infections and infestations) | 1 | 1
Gangrene (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 0 | 2
Necrotising fasciitis (Infections and infestations) | 2 | 0
Peritonitis (Infections and infestations) | 1 | 1
Pneumonia pseudomonal (Infections and infestations) | 0 | 2
Septic shock (Infections and infestations) | 1 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 1 | 1
Acinetobacter infection (Infections and infestations) | 0 | 1
Appendicitis perforated (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Cellulitis staphylococcal (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Encephalitis viral (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1
Fungal skin infection (Infections and infestations) | 1 | 0
Gallbladder empyema (Infections and infestations) | 1 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 1
Hordeolum (Infections and infestations) | 0 | 1
Infection parasitic (Infections and infestations) | 0 | 1
Intervertebral discitis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Mastoiditis (Infections and infestations) | 1 | 0
Meningitis bacterial (Infections and infestations) | 0 | 1
Nasal vestibulitis (Infections and infestations) | 1 | 0
Parasitic gastroenteritis (Infections and infestations) | 0 | 1
Parotid abscess (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Pyelonephritis chronic (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Splenic abscess (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 3 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 2
Hip fracture (Injury, poisoning and procedural complications) | 2 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 3 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 1
Patella fracture (Injury, poisoning and procedural complications) | 2 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 2
Bite (Injury, poisoning and procedural complications) | 1 | 0
Bone fissure (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Stab wound (Injury, poisoning and procedural complications) | 0 | 1
Subarachnoid haematoma (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Carbohydrate antigen 19-9 increased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Fracture delayed union (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gallbladder adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 8 | 5
Cerebral infarction (Nervous system disorders) | 4 | 8
Ischaemic stroke (Nervous system disorders) | 6 | 5
Syncope (Nervous system disorders) | 1 | 3
Cerebral ischaemia (Nervous system disorders) | 1 | 2
Transient ischaemic attack (Nervous system disorders) | 3 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Partial seizures (Nervous system disorders) | 2 | 0
Transient global amnesia (Nervous system disorders) | 0 | 2
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 1
Brain stem haemorrhage (Nervous system disorders) | 0 | 1
Brain stem infarction (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Cerebrovascular stenosis (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1
Lumbosacral radiculopathy (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Vertigo CNS origin (Nervous system disorders) | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 1 | 0
Vocal cord paresis (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 0
Delusional disorder, unspecified type (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1
Acute kidney injury (Psychiatric disorders) | 3 | 2
Chronic kidney disease (Renal and urinary disorders) | 1 | 2
Renal failure (Psychiatric disorders) | 1 | 1
Urinary retention (Psychiatric disorders) | 2 | 0
End stage renal disease (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Hypertensive nephropathy (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal injury (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Urethral polyp (Renal and urinary disorders) | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 12 | 14
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1
Pemphigus (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 7 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 3
Aortic stenosis (Vascular disorders) | 1 | 1
Hypertensive emergency (Vascular disorders) | 1 | 1
Thrombophlebitis (Vascular disorders) | 0 | 2
Aortic aneurysm (Vascular disorders) | 0 | 1
Aortic arteriosclerosis (Vascular disorders) | 0 | 1
Aortic dilatation (Vascular disorders) | 1 | 0
Diabetic vascular disorder (Vascular disorders) | 0 | 1
Embolism (Vascular disorders) | 0 | 1
Essential hypertension (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | aQIV (N=665) | Non-influenza Comparator Vaccine (N=667)
Pain (General disorders) | 106/253 | 77/193
Erythema (General disorders) | 69/218 | 69/193
Fatigue (General disorders) | 67/183 | 56/154
Headache (General disorders) | 70/161 | 53/150
Induration (General disorders) | 65/201 | 51/193
Arthralgia (General disorders) | 47/138 | 42/129
Myalgia (General disorders) | 49/134 | 39/109

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any formal publication of the study in which contribution of Seqirus personnel exceeded that of conventional monitoring will be considered as a joint publication by the investigator and the appropriate Seqirus personnel. Seqirus must be notified of any intent to publish data collected from the study and prior approval from Seqirus must be obtained prior to submission for publication.

DOCUMENTS (2):
  • Study Protocol (2017-02-06): https://cdn.clinicaltrials.gov/large-docs/21/NCT02587221/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-27): https://cdn.clinicaltrials.gov/large-docs/21/NCT02587221/SAP_001.pdf